CLINICAL TRIAL: NCT02851199
Title: The Effect of Child Position on the Results of Hyperventilation During Routine Electroencephalography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HYMC-0043-16
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study group 1 (Active Comparator): 1. A group of 15 children who will undergoe an electroencephlaography recording with 3 minutes of hyperventilation in the prone position, followed by 5 minutes of rest, then after another 5-10 minutes of recording with normal breathing. Finally the participants will performed additional 3 minutes of hyperventilation in the sitting position
  Interventions: Device: Electroencephalography
- study group 2 (Active Comparator): 2. A group of 15 children who will undergoe an electroencephlaography recording with 3 minutes of hyperventilation in the sitting position, followed by 5 minutes of rest, then after another 5-10 minutes of recording with normal breathing. . Finally the participants will performed additional 3 minutes of hyperventilation in the
  Interventions: Device: Electroencephalography

INTERVENTIONS:
Device: Electroencephalography — Electroencephalograph recording following hyperventilation in different participant's body postures

SUMMARY:
Electroencephalograhy (EEG) is used as a tool for diagnosing epilepsy/convulsions.

During the recording, especially for childen who are suspected of having abbcence epilepsy the investigators will perform an EEG recording including a provocation test of hyperventilation in order to induce epileptic discharges.

There is no clear instruction about the position of the child during performing this hyperventilation provocation.

Clinical observations showed that this provocation is more effective when it's performed in the siiting position.

No study was previously performed to investigate this issue

DETAILED DESCRIPTION:
The study will include 30 patients at the age of 4-10 years old of both sexes. after signing an informed concent, every child, suspected of having absence seizures, will undergoe an EEG recording including a provocation of hyperventilation.

The study will include two groups:

1. A group of 15 children who will undergoe an EEG recording with 3 minutes of hyperventilation in the prone position, followed by 5 minutes of rest, then after another 5-10 minutes of recording with normal breathing. Finally the participants will performed additional 3 minutes of hyperventilation in the sitting position
2. A group of 15 children who will undergoe an EEG recording with 3 minutes of hyperventilation in the sitting position, followed by 5 minutes of rest, then after another 5-10 minutes of recording with normal breathing. . Finally the participants will performed additional 3 minutes of hyperventilation in the prone position.

Participants who will not be able to perform all the steps of the study will be excluded The analysis of the study results will be performed by a specialist in pediatric neurology and pediatric epilepsy who will confirm whether the EEG recording show epileptic discharge (sharp waves, slow waves, combination of sharp and slow waves, spikes or combination of spikes and slow waves)

ELIGIBILITY:
Inclusion Criteria:

* children suspected of having absence seizures in the ages mentioned above.
* legal guardian approval

Exclusion Criteria:

* inability to perform hyperventilation
* children who have absence seizure under anti-convulsive treatment

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
epileptic discharge measurement | 1 day
  The analysis of the study results will be performed by a specialist in pediatric neurology and pediatric epilepsy who will confirm whether the EEG recording show epileptic discharge (sharp waves, slow waves, combination of sharp and slow waves, spikes or combination of spikes and slow waves)

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe medical center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Watemberg N, Farkash M, Har-Gil M, Sezer T, Goldberg-Stern H, Alehan F. Hyperventilation during routine electroencephalography: are three minutes really necessary? Pediatr Neurol. 2015 Apr;52(4):410-3. doi: 10.1016/j.pediatrneurol.2014.12.003. Epub 2014 Dec 31. PMID 25661285
- [Background] Hughes JR. Absence seizures: a review of recent reports with new concepts. Epilepsy Behav. 2009 Aug;15(4):404-12. doi: 10.1016/j.yebeh.2009.06.007. Epub 2009 Jul 24. PMID 19632158
- [Background] Ma X, Zhang Y, Yang Z, Liu X, Sun H, Qin J, Wu X, Liang J. Childhood absence epilepsy: Elctroclinical features and diagnostic criteria. Brain Dev. 2011 Feb;33(2):114-9. doi: 10.1016/j.braindev.2010.02.004. Epub 2010 Apr 7. PMID 20378290